CLINICAL TRIAL: NCT01819545
Title: Shanghai Mental Health Center
Brief Title: The Study of microRNA 107 (miRNA 107) and Beta-amyloid Precursor Protein-cleaving Enzyme 1 (BACE1) Messenger Ribonucleic Acid (mRNA) Gene Expression in Cerebrospinal Fluid and Peripheral Blood of Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government); National Natural Science Foundation of China (Other Government)
Responsible Party: Sponsor
Other Study IDs: 10ZR1425800
Record Dates: First submitted 2013-03-24; First posted 2013-03-27 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; diagnosis; MicRNA; mRNA
MeSH Terms: conditions — Alzheimer Disease; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma miRNA107 and BACE1mRNA are to be retained.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Alzheimer's disease: no intervention
- Mild cognitive impairment: no intervention
- Normal aging: no intervention

SUMMARY:
The miRNA 107 gene is increasingly appreciated to serve key functions in humans. The miRNA regulate gene expression involved in cell division, metabolism, stress response, and angiogenesis in vertebrate species. But the relationship and diagnosis capability of miRNA 107 and BACE1 mRNA gene expression in plasma and cerebrospinal fluid (CSF) of amnestic mild cognitive impairment (aMCI) and normal control is still a mystery.

DETAILED DESCRIPTION:
The Real-Time PCR was the main method in the research.

ELIGIBILITY:
Inclusion Criteria:

* Probable Alzheimer's disease (AD) was diagnosed according to the Diagnostic and Statistical Manual for Mental Disorders 4th edition (DSM-IV) criteria and the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorder's Association (NINCDS/ADRDA) criteria.
* AMCI was diagnosed based on the following criteria (Petersen et al., 2001): 1) memory complaint, preferably corroborated by a spouse or relative, 2) objective memory impairment, 3) normal general cognitive function, 4) intact activities of daily living, and 5) absence of dementia. We have amended the aMCI diagnostic criteria of the Petersen Mini-Mental State Examination (MMSE) cut-off score in order to be consistent with the low level of education in elderly Chinese people. Research (mingyuan Zhang et al, 1988) found that with the Chinese version of MMSE, AD subjects who had not been educated (NO ED) exhibited MMSE scores of <18, those with elementary school education exhibited MMSE scores of <21, and those with higher than middle school education exhibited MMSE scores of <25. In the present study, the aMCI analysis was carried out on NO ED subjects with MMSE cut-off scores of over 18, elementary school educated subjects with MMSE cut-off scores of over 21, and higher than middle school educated subject with MMSE cut-off scores of over 25.
* The cognitively-normal elderly formed the normal control (NC) group, was independently-functioning community dwellers with no neurological or psychiatric conditions.

Exclusion Criteria:

* All participants underwent a screening process that included a review of their medical history, physical and neurological examinations, laboratory tests, and MRI analysis. The clinical assessment of mild cognitive impairment or dementia included neuropsychological tests, as well as behavioral and psychiatric interviews conducted by the attending psychiatrist. AD patients recorded scores of < 4 on the Hachinski Ischemia Scale and showed no history of significant systemic or psychiatric conditions, or traumatic brain injuries that could compromise brain function.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the subjects were collected from Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine (Alzheimer's Disease and Related Disorders Center, ADRDC) and the of Shanghai Changning district, Huangpu district and Putuo district.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
plasma and CSF press of miRNA 107 and BACE1 mRNA | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Tao Wang, M.D., PhD., Principal Investigator — Department of Psychogeriatrics，Shanghai Mental Health Center
Locations (1):
- Department of Psychogeriatrics，Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang T, Shi F, Jin Y, Jiang W, Shen D, Xiao S. Abnormal Changes of Brain Cortical Anatomy and the Association with Plasma MicroRNA107 Level in Amnestic Mild Cognitive Impairment. Front Aging Neurosci. 2016 May 18;8:112. doi: 10.3389/fnagi.2016.00112. eCollection 2016. PMID 27242521
- [Derived] Wang T, Chen K, Li H, Dong S, Su N, Liu Y, Cheng Y, Dai J, Yang C, Xiao S. The feasibility of utilizing plasma MiRNA107 and BACE1 messenger RNA gene expression for clinical diagnosis of amnestic mild cognitive impairment. J Clin Psychiatry. 2015 Feb;76(2):135-41. doi: 10.4088/JCP.13m08812. PMID 25742200